CLINICAL TRIAL: NCT01196507
Title: A Prospective, Double-blind, Randomized Placebo-controlled Trial of Carvedilol for Early Primary Prophylaxis of Esophageal Varices in Cirrhosis.
Brief Title: Early Primary Prophylaxis of Esophageal Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ILBS PHT-02
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2013-12

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Tablet Carvedilol 12.5 mg BD or maximum tolerated dose
  Interventions: Drug: Carvedilol
- Placebo (Placebo Comparator): Placebo tablets 2 to 4 BD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will be administered orally at a start dose of 3.125 mg twice daily. After 1 week, this will increased if systolic blood pressure does not fall below 90 mm Hg. The patient will receive the maximum tolerated dose of carvedilol or with a maximum of 12.5 BD.
  Arms: Carvedilol
Drug: Placebo — The placebo tablets will be identical to the carvedilol tablets. First the patients will receive placebo in the dose of 1 BD. Then depending on his tolerance it will be increased to a maximum of 4 BD.
  Arms: Placebo

SUMMARY:
Patients of cirrhosis with portal hypertension aged 18 to 75 years who have small esophageal varices with or without red color signs and have not bled previously will be enrolled. After baseline evaluation, the participants will be randomized to receive either Placebo or Carvedilol 12.5 mg BD. After randomization they will be followed up for one year. The primary endpoint of the study is the the proportions of patients who develop large varices (Gd 3 or Gd 4) at 1 year in each group. The secondary endpoint are survival,reduction in HVPG,change in CTP and MELD score& adverse events.

ELIGIBILITY:
Inclusion Criteria:

- Patients of cirrhosis with portal hypertension aged 18 to 75 years who have small esophageal varices with or without red color signs and have not bled previously.

Exclusion Criteria:

* Any contra-indication to beta-blockers
* Any EVL or sclerotherapy within last 3 months
* Child Turcotte Pugh (CTP) score > 12, refractory ascites, hepatorenal syndrome
* Any past history of surgery for portal hypertension
* Significant cardio or pulmonary co-morbidity
* Any malignancy that affects survival.
* Active alcohol abuse or last intake ≤ 4 weeks to avoid possibility of ongoing alcohol hepatitis.
* Past history of surgery for portal hypertension
* Uncontrolled diabetes
* Peripheral vascular disease
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the the proportions of patients who develop large varices (Gd 3 or Gd 4) during the period of 2 year in each group. | 2 Years

SECONDARY OUTCOMES:
Survival | 2 Years
adverse effects of drugs | 2 Years
reduction in HVPG | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, MBBS, MD, DM, Principal Investigator — Institute of Liver & Biliary Sciences (ILBS)
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379